CLINICAL TRIAL: NCT04091360
Title: A Phase II, Randomised Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of Single and Repeat Doses of RPL554 Administered by Pressurised Metered Dose Inhaler in Patients With COPD
Brief Title: A Study of RPL554 Drug Administered by Metered Dose Inhaler to Treat Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RPL554-MD-201
Record Dates: First submitted 2019-06-20; First posted 2019-09-16 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: COPD
Keywords: COPD; Adults; Phase II; RPL554; Ensifentrine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Medicare Part B

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RPL554 100 mcg (Experimental): Part A: Patients receive 1 dose of either RPL554 100mcg via metered dose inhaler.
  Part B: not applicable
  Interventions: Drug: Part A: RPL554; Drug: Placebos
- RPL554 300 mcg (Experimental): Part A: Patients receive 1 dose of RPL554 300mcg via metered dose inhaler. Part B: Patients receive repeat doses of RPL554 300mcg via metered dose inhaler in crossover fashion.
  Interventions: Drug: Part A: RPL554; Drug: Placebos; Drug: Part B: RPL554
- RPL554 1000 mcg (Experimental): Part A: Patients receive 1 dose of RPL554 1000mcg via metered dose inhaler. Part B: Patients receive repeat doses of RPL554 3000mcg via metered dose inhaler in crossover fashion.
  Interventions: Drug: Part A: RPL554; Drug: Placebos; Drug: Part B: RPL554
- RPL554 3000 mcg (Experimental): Part A: Patients receive 1 dose of either RPL554 3000mcg via metered dose inhaler.
  Part B: Patients receive repeat doses of RPL554 3000mcg via metered dose inhaler in crossover fashion.
  Interventions: Drug: Part A: RPL554; Drug: Placebos; Drug: Part B: RPL554
- RPL554 6000 mcg (Experimental): Part A: Patients receive 1 dose of either RPL554 6000mcg via metered dose inhaler.
  Part B: not applicable
  Interventions: Drug: Part A: RPL554; Drug: Placebos
- RPL554 Placebo (Placebo Comparator): Part A: Patients receive 1 dose of RPL554 placebo via metered dose inhaler. Part B: Patients receive repeat doses of RPL554 placebo via metered dose inhaler in crossover fashion.
  Interventions: Drug: Part A: RPL554; Drug: Placebos

INTERVENTIONS:
Drug: Part A: RPL554 — Single dose RPL554 via metered dose inhaler.
  Other Names: Part A
Drug: Placebos — Part A: Single dose placebo via metered dose inhaler. Part B: Repeat doses of placebo via metered dose inhaler in crossover fashion. One dose administered twice daily over 7 days.
Drug: Part B: RPL554 — Part B: Repeat doses via metered dose inhaler in crossover fashion. One dose administered twice daily over 7 days.
  Other Names: Part B
  Arms: RPL554 1000 mcg; RPL554 300 mcg; RPL554 3000 mcg

SUMMARY:
The purpose of this study is to investigate 5 doses of RPL554 and placebo, administered by pressurized metered dose inhaler (pMDI), in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The study will consist of two parts. Part A is a parallel group, placebo-controlled single dose study to ascertain the Pharmacokinetics (PK) profile, safety and bronchodilator effect of a single dose of RPL554 administered via pMDI. Five of the 6 treatment arms will be double-blind and one will be single-blind (due to the different number of capsules administered). Part B is a 7-day placebo-controlled, complete block cross-over, repeat dose study to assess the bronchodilator effect of repeat doses of RPL554 delivered via pMDI.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with moderate to severe COPD, with a post bronchodilator FEV1 of 40 to 80% of predicted and FEV1/FVC ratio of ≤0.70.
* They must have a baseline increase in FEV1 of >150 mL following four puffs of salbutamol.
* They must have at least a 10 pack-year smoking history, and may be either a current or former smoker.

Exclusion Criteria:

* Patients must be clinically stable without recent COPD exacerbations or hospitalisations.
* They must not have uncontrolled disease or chronic heart failure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Respiratory Clinical Trials Ltd, London
  - Medicines Evaluation Unit Limited, Wythenshawe

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 subjects enrolled for Part A and eligible to continue into Part B.
Pre-assignment Details: Part A: 40 Patients randomized equally to receive a single dose of RPL554 (0.10, 0.30, 1, 3, or 6 mg) or matching placebo via pressurized metered dose inhaler (pMDI). Patients continued to Part B after Part A completed.
  Part B: 28 Patients continued to Part B and randomly assigned to 1 of 4 treatment sequences in a crossover design (1-week treatment periods separated by 7-10 day washout). Each sequence included twice daily RPL554 (0.30, 1, or 3 mg) or matching placebo via pMDI.
Groups:
- 0.10 mg/Part A; 0.30 mg/Part A; 1 mg/Part A; 3 mg/Part A: Part A: single dose of RPL554 via pMDI (double-blind)
- 6 mg/Part A: Part A: single dose of RPL554 via pMDI (single-blind)
- Placebo/Part A: Part A: single dose via pMDI (double-blind)
- Seq 1/Part B: Part B: 7 day, twice daily dose of RPL554 via pMDI (double-blind) complete block, cross-over.
  Seq 1= RPL554 0.30 mg / RPL554 3 mg / Placebo / RPL554 1 mg
- Seq 2/Part B: Part B: 7 day, twice daily dose of RPL554 via pMDI (double-blind) complete block, cross-over.
  Seq 2= RPL554 1 mg / Placebo / RPL554 3 mg / RPL554 0.30 mg.
- Seq 3/Part B: Part B: 7 day, twice daily dose of RPL554 via pMDI (double-blind) complete block, cross-over.
  Seq 3= RPL554 3 mg / RPL554 1 mg / RPL554 0.30 mg / Placebo.
- Seq 4/Part B: Part B: 7 day, twice daily dose of RPL554 via pMDI (double-blind) complete block, cross-over.
  Seq 4= Placebo / RPL554 0.30 mg / RPL554 1 mg / RPL554 3 mg.
Period: Part A (R, PC, PG) Single Dose
Arm/Group | 0.10 mg/Part A | 0.30 mg/Part A | 1 mg/Part A | 3 mg/Part A | 6 mg/Part A | Placebo/Part A | Seq 1/Part B | Seq 2/Part B | Seq 3/Part B | Seq 4/Part B
Started | 6 | 7 | 6 | 7 | 7 | 7 | 0 | 0 | 0 | 0
Completed | 6 | 7 | 6 | 7 | 7 | 7 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (R, PC, XO) Twice Daily for 7 Day
Arm/Group | 0.10 mg/Part A | 0.30 mg/Part A | 1 mg/Part A | 3 mg/Part A | 6 mg/Part A | Placebo/Part A | Seq 1/Part B | Seq 2/Part B | Seq 3/Part B | Seq 4/Part B
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 0.10 mg; 0.30 mg; 1 mg; 3 mg: Single dose of RPL554 via pMDI (double-blind)
- 6 mg: Single dose of RPL554 via pMDI (single-blind)
- Placebo: Single dose of placebo via pMDI (double-blind)
- Total: Total of all reporting groups
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7 | 7 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (4.92) | 71.4 (1.27) | 64.3 (7.87) | 67.1 (6.72) | 63.1 (8.71) | 64.4 (6.60) | 66.3 (6.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 3 | 2 | 3 | 16
  Male | 4 | 3 | 4 | 4 | 5 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 6 | 7 | 7 | 7 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 7 | 6 | 7 | 7 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 7 | 6 | 7 | 7 | 7 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetic Parameter AUC0-12
Description: Area under the curve from 0 to 12 hours after single dose drug administration.
Time Frame: Day 1
Population: Pharmacokinetic (PK) Analysis Set in Part A: all randomized patients who had blood sampling performed after the single dose of RPL554 and had evaluable PK parameter data. The PK Analysis Set included the 33 patients who received RPL554 in Part A but not the 7 patients in the placebo group.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7
h*pg/mL | 175 (96.7) | 611 (183) | 1550 (443) | 5860 (3120) | 9360 (8100)

2. Primary Outcome: Part A: Pharmacokinetic Parameter Cmax
Description: Pharmacokinetic Parameter Cmax after a Single Dose
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7
pg/mL | 39.4 (16.4) | 138 (40.9) | 467 (57.8) | 1520 (1050) | 2360 (1430)

3. Primary Outcome: Part A: Pharmacokinetic Parameter AUC0-t
Description: Area under the curve at maximum concentration 0-24 hrs after single dose drug administration
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 7
h*pg/mL | 208 (119) | 692 (229) | 1680 (559) | 6800 (3770) | 10800 (10100)

4. Primary Outcome: Part A: RPL554 Plasma Pharmacokinetic Parameter (Half-life)
Description: RPL554 Plasma Pharmacokinetics concentration after single dose
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg
Number analyzed (Participants) | 4 | 7 | 6 | 7 | 7
h | 6.31 (5.18) | 5.32 (3.36) | 3.47 (1.44) | 5.62 (1.7) | 4.44 (2.03)

5. Primary Outcome: Part B: Change From Baseline in Peak FEV1 (Over 4 Hours) on Day 7
Description: Change from Baseline FEV1 to Peak FEV1 (over 4 hours) after morning dosing on Day 7
Time Frame: Day 7
Population: Full Analysis Set = number of patients with at least one on treatment value who contributed to the model estimation.
Measure: Mean (Standard Deviation); unit: L
Groups:
- 0.30 mg; 1 mg; 3 mg: 7 day, twice daily dose of RPL554 via MPI (double-blind) complete block, cross-over
- Placebo: 7 day, twice daily dose of placebo via MPI (double-blind) complete block, cross-over
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22 | 23
L | 0.189 (0.1624) | 0.261 (0.1597) | 0.310 (0.1511) | -0.016 (0.1485)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.221, 95% CI 2-sided [1.163 to 1.281]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.203, 95% CI 2-sided [1.146 to 1.263]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.139, 95% CI 2-sided [1.085 to 1.195]

6. Secondary Outcome: Part A: Change From Baseline in Peak FEV1 (Over 4 Hours) After 1 Dose
Description: Change from Baseline FEV1 to Peak FEV1 (over 4 hours) After Single Dose
Time Frame: Day 1
Population: Full analysis includes patients with values at baseline and peak FEV1 (0-4h).
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7 | 7
L | 0.133 (0.1144) | 0.264 (0.1012) | 0.255 (0.0994) | 0.332 (0.2095) | 0.477 (0.1469) | 0.086 (0.0694)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.253, 95% CI 2-sided [1.151 to 1.363]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0022, ANCOVA; GeoMean Ratio = 1.146, 95% CI 2-sided [1.054 to 1.246]
Statistical Analysis 3: Comparison: 1 mg vs Placebo; Test type: Other; p = 0.0295, ANCOVA; GeoMean Ratio = 1.102, 95% CI 2-sided [1.010 to 1.202]
Statistical Analysis 4: Comparison: 0.30 mg vs Placebo; Test type: Other; p = 0.0098, ANCOVA; GeoMean Ratio = 1.129, 95% CI 2-sided [1.032 to 1.235]
Statistical Analysis 5: Comparison: 0.10 mg vs Placebo; Test type: Other; p = 0.54, ANCOVA; GeoMean Ratio = 1.028, 95% CI 2-sided [0.939 to 1.125]

7. Secondary Outcome: Part A: Change From Baseline in Average FEV1 (Over 4 Hours) After 1 Dose
Description: Change from Baseline FEV1 to Average FEV1 (over 4 hours) After Single Dose
Time Frame: Day 1
Population: Full analysis set. () () () () () ()
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7 | 7
L | 0.058 (0.0889) | 0.161 (0.0650) | 0.153 (0.0653) | 0.240 (0.1677) | 0.334 (0.1147) | -0.011 (0.0805)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.228, 95% CI 2-sided [1.142 to 1.319]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0002, ANCOVA; GeoMean Ratio = 1.155, 95% CI 2-sided [1.075 to 1.240]
Statistical Analysis 3: Comparison: 1 mg vs Placebo; Test type: Other; p = 0.0129, ANCOVA; GeoMean Ratio = 1.100, 95% CI 2-sided [1.022 to 1.184]
Statistical Analysis 4: Comparison: 0.30 mg vs Placebo; Test type: Other; p = 0.0079, ANCOVA; GeoMean Ratio = 1.112, 95% CI 2-sided [1.030 to 1.201]
Statistical Analysis 5: Comparison: 0.10 mg vs Placebo; Test type: Other; p = 0.39, ANCOVA; GeoMean Ratio = 1.033, 95% CI 2-sided [0.957 to 1.116]

8. Secondary Outcome: Part A: Change From Baseline in Average FEV1 (Over 12 Hours) After 1 Dose
Description: Change from Baseline FEV1 to Average FEV1 (over 12 hours) After Single Dose
Time Frame: Day 1
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.10 mg | 0.30 mg | 1 mg | 3 mg | 6 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 7 | 7
L | 0.018 (0.0643) | 0.061 (0.0429) | 0.010 (0.0408) | 0.121 (0.1321) | 0.190 (0.1053) | -0.031 (0.0740)
Statistical Analysis 1: Comparison: 6 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.137, 95% CI 2-sided [1.073 to 1.204]
Statistical Analysis 2: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0041, ANCOVA; GeoMean Ratio = 1.091, 95% CI 2-sided [1.030 to 1.155]
Statistical Analysis 3: Comparison: 1 mg vs Placebo; Test type: Other; p = 0.53, ANCOVA; GeoMean Ratio = 1.019, 95% CI 2-sided [0.960 to 1.081]

9. Secondary Outcome: Part A: Safety and Tolerability / Hematology Safety Assessments
Description: Number of patients with treatment-emergent hematology abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

10. Secondary Outcome: Part A: Safety and Tolerability / Blood Chemistry Safety Assessments: Number of Patients With Treatment-emergent Blood Chemistry Abnormal Laboratory Assessments
Description: Number of patients with treatment-emergent blood chemistry abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

11. Secondary Outcome: Part A: Safety and Tolerability / Urinalysis Safety Assessments: Number of Patients With Treatment-emergent Urinalysis Abnormal Laboratory Assessments
Description: Number of patients with treatment-emergent urinalysis abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

12. Secondary Outcome: Part A: Safety and Tolerability / Supine Vitals Signs - Pulse Rate
Description: Number of patients with treatment-emergent abnormal vital signs (pulse rate in bpm)
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

13. Secondary Outcome: Part A: Safety and Tolerability / Supine Vitals Signs - Blood Pressure
Description: Number of patients with treatment-emergent abnormal vital signs (blood pressure in mm Hg)
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

14. Secondary Outcome: Part A: Safety and Tolerability / ECG - QTcF
Description: Number of patients with treatment-emergent abnormal ECG parameters, QTcF in msec
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

15. Secondary Outcome: Part A: Safety and Tolerability / ECG - Heart Rate
Description: Number of patients with treatment-emergent abnormal ECG parameters, heart rate in bpm
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

16. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 4 Hrs) After 7 Days
Description: Change from baseline in average FEV1 (over 4 hours) on Day 7 after morning dose
Time Frame: Day 7
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22 | 23
L | 0.083 (0.1223) | 0.161 (0.1686) | 0.206 (0.1470) | -0.095 (0.1702)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.210, 95% CI 2-sided [1.153 to 1.270]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.193, 95% CI 2-sided [1.136 to 1.252]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.124, 95% CI 2-sided [1.071 to 1.179]

17. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 12 Hours) After 7 Days
Description: Change from baseline FEV1 in average FEV1 (over 12 hours) on Day 7 after morning dose
Time Frame: Day 7
Population: Full analysis Set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22 | 23
L | 0.008 (0.1421) | 0.075 (0.1472) | 0.085 (0.1411) | -0.112 (0.1662)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.139, 95% CI 2-sided [1.087 to 1.194]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.142, 95% CI 2-sided [1.089 to 1.197]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p = 0.0018, ANCOVA; GeoMean Ratio = 1.080, 95% CI 2-sided [1.031 to 1.132]

18. Secondary Outcome: Part B: Change From Baseline in Trough FEV1 After 7 Days
Description: Change from Baseline FEV1 to Morning Trough FEV1 on Day 7 after morning dose
Time Frame: Day 7
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 22 | 22 | 23
L | -0.051 (0.1254) | -0.017 (0.1783) | 0.013 (0.1631) | -0.097 (0.1389)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p = 0.0066, ANCOVA; GeoMean Ratio = 1.080, 95% CI 2-sided [1.022 to 1.140]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p = 0.0115, ANCOVA; GeoMean Ratio = 1.074, 95% CI 2-sided [1.017 to 1.134]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p = 0.18, ANCOVA; GeoMean Ratio = 1.037, 95% CI 2-sided [0.982 to 1.096]

19. Secondary Outcome: Part B: Change From Baseline in Peak FEV1 (Over 4 Hours) After 1st Dose
Description: Change from baseline FEV1 in peak FEV1 (over 4 hours) after first dose
Time Frame: Day 1
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
L | 0.253 (0.0772) | 0.311 (0.1532) | 0.337 (0.1108) | 0.079 (0.0914)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.162, 95% CI 2-sided [1.122 to 1.203]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.150, 95% CI 2-sided [1.111 to 1.190]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.112, 95% CI 2-sided [1.074 to 1.152]

20. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 4 Hours) After 1st Dose
Description: Change from baseline FEV1 in average FEV1 (over 4 hours) on Day 1
Time Frame: Day 1
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
L | 0.144 (0.0762) | 0.204 (0.1162) | 0.224 (0.0905) | -0.017 (0.1284)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.157, 95% CI 2-sided [1.119 to 1.196]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.147, 95% CI 2-sided [1.110 to 1.186]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.105, 95% CI 2-sided [1.068 to 1.142]

21. Secondary Outcome: Part B: Change From Baseline in Average FEV1 (Over 12 Hours) After 1st Dose
Description: Change from baseline FEV1 in average FEV1 (over 12 hours) on Day 1
Time Frame: Day 1
Population: number of patients with at least one on treatment value who contributed to the model.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 0.30 mg | 1 mg | 3 mg | Placebo
Number analyzed (Participants) | 22 | 23 | 22 | 23
L | 0.047 (0.0914) | 0.102 (0.1306) | 0.085 (0.0659) | -0.058 (0.1444)
Statistical Analysis 1: Comparison: 3 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.098, 95% CI 2-sided [1.059 to 1.137]
Statistical Analysis 2: Comparison: 1 mg vs Placebo; Test type: Other; p < 0.0001, ANCOVA; GeoMean Ratio = 1.111, 95% CI 2-sided [1.072 to 1.150]
Statistical Analysis 3: Comparison: 0.30 mg vs Placebo; Test type: Other; p = 0.0003, ANCOVA; GeoMean Ratio = 1.070, 5% CI 2-sided [1.033 to 1.109]

22. Secondary Outcome: Part B: RPL554 Plasma Pharmacokinetic Parameter (Onset of Action)
Description: Determination of onset of action (>10% increase in FEV1 from pre- to post-first dose, censored at 120 minutes) on Day 1
Time Frame: Day 1
Population: Patients with onset of action
Measure: Median (Full Range); unit: mins
Arm/Group | 0.30 mg | 1 mg | 3 mg
Number analyzed (Participants) | 18 | 19 | 22
mins | 37.0 [3 to 120] | 27.5 [5 to 120] | 19.0 [5 to 91]
Statistical Analysis 1: Comparison: 1 mg vs 3 mg; Test type: Other; p = 0.47, Hodges-Lehmann; Median Difference (Final Values) = 8.5
Statistical Analysis 2: Comparison: 0.30 mg vs 3 mg; Test type: Other; p = 0.0059, Hodges-Lehmann; Mean Difference (Final Values) = 18.0

23. Secondary Outcome: Part B: Safety and Tolerability / Hematology Safety Assessments
Description: Number of patients with treatment-emergent hematology abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

24. Secondary Outcome: Part B: Safety and Tolerability / Blood Chemistry Safety Assessments
Description: Number of patients with treatment-emergent blood chemistry abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

25. Secondary Outcome: Part B: Safety and Tolerability / Urinalysis Safety Assessments
Description: Number of patients with treatment-emergent urinalysis abnormal laboratory assessments
Time Frame: 1 day
Reporting Status: Not Posted

26. Secondary Outcome: Part B: Safety and Tolerability / Supine Vital Signs - Pulse Rate
Description: Number of patients with treatment-emergent abnormal vital signs (pulse rate in bpm)
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

27. Secondary Outcome: Part B: Safety and Tolerability / Supine Vital Signs - Blood Pressure
Description: Number of patients with treatment-emergent abnormal vital signs (blood pressure in mm Hg)
Time Frame: Start of treatment to day 1
Reporting Status: Not Posted

28. Secondary Outcome: Part B: Safety and Tolerability / ECG - QTcF
Description: Number of patients with treatment-emergent abnormal ECG parameters, QTcF in msec
Time Frame: Start of treatment to day 70
Reporting Status: Not Posted

29. Secondary Outcome: Part B: Safety and Tolerability / ECG - Heart Rate
Description: Number of patients with treatment-emergent abnormal ECG parameters, heart rate in bpm
Time Frame: Start of treatment to day 70
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Part A: 24 hours. Part B: Approximately 70 days
Groups:
- Part B/0.30 mg; Part B/1 mg; Part B/3 mg: Part B: 7 day, twice daily dose of RPL554 via pMDI (double-blind) complete block, cross-over.
- Part B/Placebo: Part B: 7 day, twice daily dose of placebo via pMDI (double-blind) complete block, cross-over.
Arm/Group | 0.10 mg/Part A | 0.30 mg/Part A | 1 mg/Part A | 3 mg/Part A | 6 mg/Part A | Placebo/Part A | Part B/0.30 mg | Part B/1 mg | Part B/3 mg | Part B/Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/7 | 0/7 | 0/7 | 0/24 | 0/23 | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/7 | 0/7 | 0/7 | 0/24 | 0/23 | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 2/6 | 1/7 | 1/6 | 2/7 | 4/7 | 2/7 | 3/24 | 4/23 | 2/23 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.10 mg/Part A (N=6) | 0.30 mg/Part A (N=7) | 1 mg/Part A (N=6) | 3 mg/Part A (N=7) | 6 mg/Part A (N=7) | Placebo/Part A (N=7) | Part B/0.30 mg (N=24) | Part B/1 mg (N=23) | Part B/3 mg (N=23) | Part B/Placebo (N=25)
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT04091360/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04091360/SAP_001.pdf